CLINICAL TRIAL: NCT04469946
Title: Short-Term Pediatric Acclimatization to Adaptive Hearing Aid Technology
Brief Title: Hearing Aid Noise Reduction in Pediatric Users Pilot Study (Oticon Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-5953-2
Record Dates: First submitted 2020-06-21; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Hearing Impairment; Sensorineural Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Pediatric hearing aid users (6 to 12 years old) participated in an intervention trial of a hearing aid with an integrated directionality and noise reduction program. Pre- to post-comparison measures were obtained after two months of intervention use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exploratory (Experimental): Participants were fit with Oticon OPN™ behind-the-ear hearing aids with the OpenSound Navigator algorithm enabled. Pre-intervention measures were obtained within one week of the hearing aid fit and post-intervention measures were obtained after two months of daily hearing aid use.
  Interventions: Device: Oticon OpenSound Navigator speech enhancement algorithm

INTERVENTIONS:
Device: Oticon OpenSound Navigator speech enhancement algorithm — OpenSound Navigator (OSN) is a speech enhancement algorithm developed by Oticon. The feature is built in Oticon's current OPN™ hearing aid platform and can be adjusted and disabled in the programming. It is designed to automatically enhance speech while reducing unwanted background noise to improve communication for the user.
  Other Names: OSN

SUMMARY:
The purpose of this study is to evaluate the efficacy of OpenSound Navigator (OSN), a hearing aid speech-enhancement algorithm developed by Oticon, as treatment for pediatric hearing aid users. The study used a within-subjects design with pre- and post-comparisons involving fifteen pediatric (ages 6-12) patients with symmetrical sensorineural hearing losses ranging from the mild to moderately-severe degree. All participants were fit with bilateral Oticon OPN™ behind-the-ear hearing aids set with the OSN algorithm enabled. The investigators evaluated hearing aid benefit through word recognition in noise (behavioral testing) and everyday hearing/listening abilities (parental/legal guardian reported) within one week of the hearing aid fitting (pre-intervention) and two months post fitting (post-intervention).

DETAILED DESCRIPTION:
OpenSound Navigator (OSN) is a speech enhancement hearing aid algorithm developed by Oticon that utilizes an adaptive directional microphone system with an automatic gain control noise reduction program. This hearing aid feature is intended for adult hearing aid users and its potential benefits of speech, vocabulary and listening development in pediatric users has not been investigated. Here the investigators aim to evaluate the efficacy of OSN programming in pediatric hearing aid users (6-12 years of age) diagnosed with a symmetrical sensorineural hearing loss in the mild to moderately-severe range. The investigators used a within-subjects study design with pre- and post-comparisons. All participants were fit with bilateral Oticon OPN™ behind-the-ear hearing aids with the OSN feature enabled. Participants will undergo standard audiometric diagnostic testing and will be fit with the hearing aids by a licensed clinical audiologist. Participants are required to wear the hearing aids full time (at least 6 hours per day average) during the duration of the study. The evaluation measures will include speech recognition testing in controlled background noise and the Speech, Spatial and Qualities of Hearing Scale questionnaire (completed by parents/legal guardian). Testing will be performed within a week of the hearing aid fitting (pre-intervention) and two months post fitting (post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* children ages 6 to 12 years
* English as the primary home language
* positive for bilateral symmetrical mild to moderately-severe sensorineural hearing loss
* currently using hearing aids that were dispensed at least 18 months prior to enrollment of the study
* negative for major cognitive handicap or developmental delay that would prevent or restrict participation, as determined by the PI or designee
* negative for learning disability, for example attention-deficit/hyperactivity disorder, as determined by the PI or designee
* negative for serious neurological or psychiatric disease that would prevent or restrict participation, as determined by the PI or designee
* informed consent of parent/guardian
* assent of participating child if aged 11 years and over
* standard MRI inclusion criteria as set by the Cincinnati Children's Hospital Medical Center department of Radiology
* not currently pregnant or breast feeding
* willingness and ability of the participant and/or the participant's caregiver to comply with study requirements
* no history of medical neglect of caregiver

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Word Recognition in Noise Abilities | 2 months
  Aided speech perception in noise was evaluated using a novel word recognition in noise test. Recorded target word intensity was fixed at 65 decibels (dB) sound pressure level (SPL) with an adaptive noise level set at an initial level of 55 dB SPL. Participants were instructed to keep their head still, listen closely to the target word and repeat the word back. If the repeated word was correct, the noise level increased by 4 dB, if incorrect, the noise reduced by 4 dB. After the second reversal, the adaptive noise level changed to 2 dB increments. This continued for six more noise level reversals for an overall signal-to-noise ratio (SNR) threshold calculation. The final threshold score indicates the estimated SNR level in which the participant correctly recognizes monosyllabic words 50% of the time (SNR-50). This test was performed within a week of hearing aid fitting and again after two months.
Word Recognition in Quiet Abilities | 2 months
  Aided speech perception in quiet was evaluated within a week of hearing aid fitting and again after two months. Recorded sentences were presented at 50 dB SPL, and scoring was based on accuracy of each recited word.
Memory | 2 months
  Long-term vocabulary memory and episodic memory were evaluated using subtests from the standardized NIH Tool Box test. Subtests included the Picture Vocabulary test and the Picture Sequence Memory Test. Tests produced a standardized age-adjusted numeric score. Testing was completed within a week of hearing aid fitting and again after two months.
Executive Function | 2 months
  Executive function was evaluated using subtests from the standardized NIH Tool Box test. Subtests included the Flanker Inhibitory Control and Attention test and and the Dimensional Change Card Sort test. Tests produced a standardized age-adjusted numeric score. Testing was completed within a week of hearing aid fitting and again after two months.
Mathematic Academic Performance | 2 months
  Mathematic skills were evaluated using a standardized battery called the Woodcock-Johnson IV Test of Achievement (WJ-IV). Subtests included Applied Problems and Calculation. Tests produced a standardized age-adjusted numeric score. Testing was completed within a week of hearing aid fitting and again after two months.
Academic Language Performance | 2 months
  Language skills were evaluated using WJ-IV. Subtests included Letter-Word Identification and Passage Comprehension. Tests produced a standardized age-adjusted numeric score. Testing was completed within a week of hearing aid fitting and again after two months.

SECONDARY OUTCOMES:
Speech, Spatial Qualities of Hearing Scale (SSQ) Scores | 2 months
  Speech, Spatial and Qualities of Hearing Scale (SSQ), a survey utilizing an ordinal scale specifically measuring hearing aid benefit with regard to speech understanding, spatial awareness, perceptual quality of sound, and conversation, was completed by parents/legal guardian within a week of the hearing aid fitting and after wearing the study hearing aids for two months. There are 4 survey sections. Section A: Speech has 8 questions, Section B: Spatial Hearing has 5 questions, Section C: Qualities of Hearing has 8 questions and Section D: Conversational Uses of Hearing has 5 questions. Each question uses a scale ranging from 0 (poorest possible outcome) to 100 (best possible outcome). Each section calculates an average score across the corresponding questions for a total of 4 individual scores.
Glasgow Hearing Aid Benefit Profile Scores | 2 months
  Glasgow Hearing Aid Benefit Profile, a survey utilizing an ordinal scale with regard to perceived hearing aid benefit was completed by parents/legal guardians within a week of the hearing aid fit and after two months of hearing aid use. It includes 24 questions assessing change in hearing disability, handicap, hearing aid use, benefit and satisfaction and residual (aided) disability relative to the benefit of their previous hearing aids. Each question uses a scale ranging from -100 (reduced benefit) to +100 (increased benefit) with all questions averaged to make a final numeric score.

CONTACTS AND LOCATIONS:
Overall Officials: David R Moore, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No